CLINICAL TRIAL: NCT00069602
Title: DirecNet Pilot Study to Assess the Accuracy of Continuous Glucose Monitors in Normal Children
Brief Title: Assessing Continuous Glucose Monitors in Healthy Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DirecNet 002; HD041890; HD041919-01; HD041908-01; HD041906-01; HD041918-01; HD041915
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus
Keywords: Continuous Glucose Monitoring Devices; Blood glucose profiles in normal children; Blood glucose profiles in non-diabetic children
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring System (CGMS)
Device: GlucoWatch G2TM Biographer (GW2B)

SUMMARY:
Continuous glucose monitors may be useful in the treatment of children with Type 1 diabetes mellitus. The purpose of this study was to determine whether two FDA-approved continuous glucose monitors, the Continuous Glucose Monitoring System (CGMS) and the GlucoWatch G2TM Biographer (GW2B), are sufficiently accurate to use in future studies to characterize glucose levels in children.

DETAILED DESCRIPTION:
The characterization of glucose levels in healthy children during day and nighttime is critical to the interpretation of glucose levels in diseases such as diabetes. This study was conducted by the DirecNet Study Group to determine whether two FDA-approved continuous glucose monitors are sufficiently accurate.

The study was conducted at five clinical centers and enrolled approximately 20 healthy children (ages 7 to 17 years old) who did not have Type 1 or Type 2 diabetes nor a history of the disease in their immediate families. Each participant was hospitalized for approximately 26 hours to assess the accuracy of the continuous glucose monitors compared with serum glucose determinations.

ELIGIBILITY:
Inclusion Criteria

* Weight >= 16.0 kg (35 lbs)
* Body mass index between the 10th to 90th percentile for age and sex
* HbA1c within normal limits
* Hematocrit within normal limits

Exclusion Criteria

* History of diabetes
* History of positive islet cell antibody testing
* Family history of Type 1 or Type 2 diabetes in a sibling or parent
* Medication use of any type in the 7 days prior to study entry
* Skin abnormalities contraindicating device use

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20
Dates: Start 2002-08; Study Completion 2002-11

PRIMARY OUTCOMES:
Accuracy of the GlucoWatch G2 Biographer and CGMS sensors

CONTACTS AND LOCATIONS:
Overall Officials: William V. Tamborlane, MD, Study Chair — Yale University
Locations (6):
- United States (6):
  - Division of Pediatric Endocrinology and Diabetes, Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Denver, Colorado
  - Department of Pediatrics, Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jaeb Center for Health Research, Tampa, Florida
  - Department of Pediatrics, University of Iowa Carver College of Medicine, Iowa City, Iowa

REFERENCES:
- [Background] Mauras N, Beck R, Ruedy K, Booth A, Weinzimer S, and the Diabetes Research in Children Network (DirecNet) Study Group. The Physiological Variations of Plasma Glucose Concentrations in Healthy, Non-Diabetic Children: Use of Continuous Glucose Sensors. Pediatr Res 2003 Apr;53(4Pt 2):1A-669A
- [Background] Weinzimer S, Beck R, Ruedy K, Booth A, Boland E, and the Diabetes Research in Children Network (DirecNet) Study Group. Mealtime Glycemic Excursions in Pediatric Subjects with Type 1 Diabetes Mellitus (T1DM): The DirecNet Experience.Pediatr Res 2003 Apr;53(4Pt2):1A-669A
- [Background] Tsalikian E, Beck R, Ruedy K, Booth A, Tansey M, and the Diabetes Research in Children Network (DirecNet) Study Group. Glycemic Pattern of Insulin Induced Hypoglycemia in Pediatric Subjects with Type 1 Diabetes Mellitus (T1DM): The DirecNet Experience. Pediatr Res 2003 Apr;53(4Pt2):1A-669A
- [Background] Buckingham B, Beck R, Tamborlane W, Ruedy K, Boland E, Chase P, Wysocki T, Tsalikian E, Wilson D, Mauras N, Weinzimer D, Tansey M, Fiallo-Scharer R, Booth A, Kollman C, and the Diabetes Research In Children Network (DirecNet) Study Group. Diabetes Research in Children Network (DirecNet) Accuracy Study of the Continuous Glucose Monitoring System (CGMS) and GlucoWatch® G2™ Biographer (GWB) in Children with Type 1 Diabetes-A CRC-based Study. Diabetes 2003 Jun;52 Suppl 1:A36.
- [Background] Wilson D, Buckingham B, Beck R, Ruedy K, Kollman C, Tsalikian E, Wysocki T, Weinzimer S, Chase P, and the Diabetes Research in Children Network (DirecNet) Study Group. A 5-center CRC-based Study of the Accuracy of the GlucoWatch®G2™ Biographer in Children and Adolescents with Type 1 Diabetes. Diabetes 2003 Jun;52 Suppl 1:A101.
- [Background] Boland E, Weinzimer S, Beck R, Ruedy K, Kollman C, Buckingham B, Chase P, Tansey M, Mauras N, and the Diabetes Research In Children Network (DirecNet) Study Group. Performance of the Medtronic MiniMed Continuous Glucose Monitoring System (CGMS) in Children with T1DM in the DirecNet Accuracy Study. Diabetes 2003 Jun;52 Suppl 1:A90.
- [Background] Fiallo-Scharer R, Chase P, Beck R, Ruedy K, Booth A, Wysocki T, Boland E, Buckingham B, Tsalikian E, and the Diabetes Research In Children Network (DirecNet) Study Group. Performance of the One Touch Ultra at Different Glucose Levels in Three Age Groups of Children with T1DM in the CRC-DirecNet Accuracy Study. Diabetes 2003 Jun;52 Suppl 1:A562.
- [Background] Mauras N, Beck RW, Ruedy KJ, Kollman C, Tamborlane WV, Chase HP, Buckingham BA, Tsalikian E, Weinzimer S, Booth AD, Xing D; Diabetes Research in Children Network (DirecNet) Accuracy Study. Lack of accuracy of continuous glucose sensors in healthy, nondiabetic children: results of the Diabetes Research in Children Network (DirecNet) accuracy study. J Pediatr. 2004 Jun;144(6):770-5. doi: 10.1016/j.jpeds.2004.03.042. PMID 15192625